CLINICAL TRIAL: NCT01301716
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of GDC-0980 in Combination With Either Paclitaxel and Carboplatin (With or Without Bevacizumab) or Pemetrexed and Cisplatin in Patients With Solid Tumors
Brief Title: A Study of the Safety and Pharmacology of GDC-0980 in Combination With Either Paclitaxel and Carboplatin (With or Without Bevacizumab) or Pemetrexed and Cisplatin in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIM4946g; GO01336 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers
MeSH Terms: interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one; Bevacizumab; Carboplatin; Cisplatin; Paclitaxel; Pemetrexed

ARMS (3):
- A (Experimental)
  Interventions: Drug: GDC-0980; Drug: carboplatin; Drug: paclitaxel
- B (Experimental)
  Interventions: Drug: GDC-0980; Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- C (Experimental)
  Interventions: Drug: GDC-0980; Drug: cisplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: GDC-0980 — Oral escalating dose
Drug: bevacizumab — Intravenous repeating dose
  Arms: B
Drug: carboplatin — Intravenous repeating dose
  Arms: A; B
Drug: cisplatin — intravenous repeating dose
  Arms: C
Drug: paclitaxel — Intravenous repeating dose
  Arms: A; B
Drug: pemetrexed — intravenous repeating dose
  Arms: C

SUMMARY:
This is an open-label, multicenter, Phase Ib dose-escalation study to assess the safety, tolerability, and pharmacokinetics of GDC-0980 administered with either paclitaxel and carboplatin (with or without bevacizumab) or pemetrexed and cisplatin to patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable, locally advanced, or metastatic solid malignancy
* Adequate hematologic and end organ function
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement to use an effective form of contraception and to continue its use for the duration of the study
* Measurable disease per RECIST (Response Evaluable Criteria in Solid Tumors), with the exception of prostate cancer (two rising PSA Levels that meet the criteria of progression per PSA Working Group) and ovarian cancer (two rising CA-125 levels greater than the ULN)

Exclusion Criteria:

* Current dyspnea at rest due to complications of advanced malignancy, or other conditions requiring continuous supplemental oxygen
* Uncontrolled hypomagnesemia or hypokalemia
* History of Grade >= 3 fasting hyperglycemia
* Any condition requiring full-dose anticoagulants
* Known HIV infection
* Known untreated or active central nervous system (CNS) metastases
* Pregnancy, lactation, or breastfeeding
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of study treatment or anticipation of need for major surgical procedure during the course of the study
* For Arm B: Conditions that preclude the use of bevacizumab
* For Arm C: Conditions that preclude the use of pemetrexed or cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of study treatment or initiation of new anti-cancer therapy, whichever comes first
Incidence of dose limiting toxicities (DLTs) | Up to 21 days from Last Patient In (LPI) in Stage 1 of study
Nature of adverse events | Up to 30 days after last dose of study treatment or initiation of new anti-cancer therapy, whichever comes first
Nature of dose limiting toxicities (DLTs) | Up to 21 days from Last Patient In (LPI) in Stage 1 of study
Severity of adverse events | Up to 30 days after last dose of study treatment

SECONDARY OUTCOMES:
Total exposure | Up to 32 months or early study discontinuation
Maximum plasma concentration | Up to 32 months or early study discontinuation
Time to maximum observed plasma concentration | Up to 32 months or early study discontinuation
Plasma half-life | Up to 32 months or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (3):
  - Los Angeles, California
  - Tampa, Florida
  - Boston, Massachusetts
- Madrid, Madrid, Spain